CLINICAL TRIAL: NCT00955175
Title: Radiation Dose Escalation For Non-Small Cell Lung Cancer Using Hypofractionated 3-Dimensional Conformal Radiation Therapy
Brief Title: Hypofractionated 3-Dimensional Radiation Therapy in Treating Patients With Newly Diagnosed Stage I, Stage II, or Stage III Non-Small Cell Lung Cancer. ICORG 99-09
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 99-09 ICORG; ICORG-99-09; EU-20922
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

ARMS (3):
- Group 1 (Experimental): Patients undergo hypofractionated 3-dimensional conformal radiotherapy 5 days a week for 24 fractions (total of 72 Gy).
  Interventions: Radiation: hypofractionated radiation therapy
- Group 2 (Experimental): Patients undergo hypofractionated 3-dimensional conformal radiotherapy 5 days a week for 22 fractions (total of 66 Gy).
  Interventions: Radiation: hypofractionated radiation therapy
- Group 3 (Experimental): Patients undergo hypofractionated 3-dimensional conformal radiotherapy 5 days a week for 20 fractions (total of 60 Gy).
  Interventions: Radiation: hypofractionated radiation therapy

INTERVENTIONS:
Radiation: hypofractionated radiation therapy — Given 5 days a week for 20, 22, or 24 fractions

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high dose of radiation directly to the tumor over a shorter period of time may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: This phase II trial is studying the side effects of hypofractionated 3-dimensional radiation therapy and to see how well it works in treating patients with newly diagnosed stage I, stage II, or stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the acute and long-term radio-induced toxicity (any organ) of hypofractionated 3-dimensional conformal radiotherapy in patients with newly diagnosed stage I-III non-small cell lung cancer.

Secondary

* To assess the radiological tumor response rate at 3 months after completion of radiotherapy.
* To assess the actuarial freedom from thoracic progression rate.

OUTLINE: Patients are stratified according to combined lung volume at 25 Gy (≤ 30% vs > 30%). Patients are assigned to 1 of 3 treatment groups.

* Group 1: Patients undergo hypofractionated 3-dimensional conformal radiotherapy 5 days a week for 24 fractions (total of 72 Gy).
* Group 2: Patients undergo hypofractionated 3-dimensional conformal radiotherapy 5 days a week for 22 fractions (total of 66 Gy).
* Group 3: Patients undergo hypofractionated 3-dimensional conformal radiotherapy 5 days a week for 20 fractions (total of 60 Gy).

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed newly diagnosed non-small cell lung cancer meeting 1 of the following stage criteria:

  * Stage I or II disease

    * Medically inoperable or patient refused surgery
  * Stage IIIA or IIIB disease (no pleural effusions)
* Radiation dose parameters must satisfy the required study dose-volume constraints

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Weight loss ≤ 10% within 3 months before diagnosis
* No other malignancy within the past 5 years, except nonmelanoma skin cancer
* No clinically significant cardiovascular disease (e.g., hypertension [blood pressure > 150/100 mm Hg], myocardial infarction or stroke within the past 6 months, or unstable angina)

PRIOR CONCURRENT THERAPY:

* No concurrent chemotherapy

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2000-11; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Acute radio-induced toxicity as assessed by the RTOG/EORTC acute toxicity grading system weekly during radiotherapy | weekly during radiotherapy
Long-term radio-induced toxicity as assessed by the long-term RTOG/EORTC and SWOG (lung) grading system every 3 months for 2 years and then every 6 months thereafter | every 3 months for 2 years and then every 6 months thereafter

SECONDARY OUTCOMES:
Tumor response rate (according to WHO response criteria) as assessed by CT scan at 3 months after completion of radiotherapy | at 3 months after completion of radiotherapy
Actuarial freedom from thoracic progression rate | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Thirion, MD, Principal Investigator — Saint Luke's Hospital
Locations (1):
- Saint Luke's Hospital, Dublin, Ireland